CLINICAL TRIAL: NCT03506061
Title: iPS Cell Response to CFTR Modulators: Study of Trikafta in CF Patients Carrying Partial Function Mutations or N1303K CFTR
Brief Title: Trikafta in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cystic Fibrosis Foundation (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Eric Sorscher, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00108656; 300001205 (Other: University of Alabama); R01HL139876 (NIH)
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor; tezacaftor; elexacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Substudy 1 - Participants With Evidence of Partial Function (Experimental): Participants with CF with evidence of partial function (sweat chloride < 80 milliequivalents per liter (mEq/L) or pancreatic sufficiency) will receive Trikafta for 28 days.
  Interventions: Drug: Trikafta
- Substudy 2 - Participants who Encode the N1303K Variant (Experimental): Participants with CF who encode the N1303K variant will receive Trikafta for 28 days.
  Interventions: Drug: Trikafta

INTERVENTIONS:
Drug: Trikafta — Participants will take Trikafta which is a combination tablet comprised of 100 milligrams (mg) of elexacaftor, 50 mg of tezacaftor and 75 mg of ivacaftor (2 tablets taken in the morning), and 150 mg of ivacaftor taken in the evening.
  Other Names: ivacaftor; tezacaftor; elexacaftor

SUMMARY:
This clinical study will enroll 42 participants without the F508del mutation, carrying partial function or N1303K mutations not approved for Trikafta, and who are not expected to be approved for CFTR modulator treatment in the immediate future. Each participant will be given Trikafta for approximately four weeks. The study researchers will monitor clinical endpoints that include forced expiratory volume (FEV1) and sweat chloride. Additionally, the researchers will obtain skin biopsy material and/or blood sample from each subject so that induced pluripotent stem (iPS) cells can be modified into airway cell monolayers and tested for response to Trikafta. In this way, the study will evaluate an emerging and readily accessible in vitro endpoint as a predictor of clinical response. This study will serve as a pilot/test case for other clinical protocols relevant to patients with rare CFTR variants who do not currently receive modulator therapies.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is a life threatening genetic disorder resulting from mutations found in the gene known as the cystic fibrosis transmembrane conductance regulator (CFTR). Defects in this gene prevent correct chloride and bicarbonate transport in and out of cells. It has become increasingly important to develop new in vitro model systems capable of predicting in vivo clinical effectiveness of modulator therapy among patients with CF. This objective represents a significant and unmet need for advancing personalized therapeutics in the disease.

Trikafta is currently approved for patients with CF carrying at least one copy of the common F508del variant and over 250 other CFTR abnormalities. Because approximately 90% of CF patients in the United States meet these criteria, pharmacotherapies (Trikafta in particular) are now available to a sizable majority of those with the disease. However, thousands of patients harboring relatively common variants will remain without effective drug therapy. Others with ultra-rare or private CFTR mutations have forms of the disease that are very likely to benefit from available drugs, but do not have access to these therapies. It has been estimated that over 1,000 CFTR mutations are represented by less than 5 patients each. Establishing processes so that individuals with very rare and/or poorly characterized alleles can gain access to effective modulator treatment remains one of the predominant challenges in the field.

This clinical study will enroll 42 participants without the F508del mutation, carrying partial function or N1303K mutations not approved for Trikafta. Substudy 1 will comprise an open-label, two center trial of orally administered elexacaftor, tezacaftor and ivacaftor (Trikafta) that will enroll 22 patients with rare/orphan genotypes. Substudy 2 will enroll 20 participants who encode the N1303K variant as emblematic of a mutation not approved for Trikafta, but are likely to respond to the treatment.

Each participant will have clinical and/or preclinical evidence that Trikafta should offer benefit, and each will be given Trikafta for approximately four weeks. The researchers will monitor clinical endpoints that include FEV1, sweat chloride, quality of life, and weight. The study will differentiate iPS cells from each subject to generate airway epithelial monolayers that can be tested for response to Trikafta. This trial will serve as a pilot/test case for other clinical protocols relevant to patients with rare CFTR variants and evidence of residual function who do not have an approved modulator therapy, due to rarity of their mutation. It is hypothesized that a correlation will be established between in vitro Trikafta responsiveness of iPS cells and in vivo benefit (FEV1) in patients, and provide a tool for utilizing iPS cells to identify rare CF patient populations most suitable for cystic fibrosis modulator therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form or assent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female age ≥12
* A clinical diagnosis of CF or CFTR-related disease and either: 1) evidence for a partial function mutation not currently covered or likely to be covered for treatment with a CFTR modulator (Substudy 1), or 2) N1303K CFTR and a minimal function mutation (Substudy 2)
* Sweat Chloride < 80 mmol/L and/or pancreatic sufficiency (no exogenous pancreatic enzyme supplement therapy) or carrying the N1303K CFTR variant
* Able to perform spirometry meeting American Thoracic Society (ATS) criteria for acceptability and repeatability
* Clinically stable in the past 4 weeks with no evidence of CF exacerbation (prior to screening and study Day 1)
* Willingness to use at least one form of acceptable birth control including abstinence or condom with spermicide. This will include birth control for at least one month prior to screening and agreement to use such a method during study participation for an additional four weeks after the last administration of study drug
* Ability to take Trikafta
* Agreement to adhere to all current medical therapies as designated by the CF care center physician

Exclusion Criteria:

* Documented history of drug or alcohol abuse within the last year
* Subjects should not have a pulmonary exacerbation or changes in therapy for pulmonary disease in the 4 weeks prior to screening
* Listed for lung or liver transplant at the time of screening
* Cirrhosis or elevated liver transaminases > 3 times the upper limit of normal
* Pregnant or breastfeeding
* Inhibitors or inducers of CYP3A4, including certain herbal medications and grapefruit/grapefruit juice, or other medicines known to negatively influence Trikafta administration
* History of solid organ transplant
* Active therapy for non-tuberculosis mycobacterial infection or any plan to initiate non-tuberculosis mycobacterial therapies during the study period
* Known allergy to Trikafta
* Treatment in the last 6 months with an approved CFTR modulator
* Any other condition that in the opinion of the lead investigators might confound results of the study or pose an additional risk from administering study drug
* Treatment with another investigational drug or other intervention within one month prior to enrollment, throughout the duration of study participation, and for an additional four weeks following final drug administration
* Evidence of cataract/lens opacity determined to be clinically significant by an ophthalmologist at or within 3 months prior to the Screening Visit

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sorscher, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - University of Alabama Cystic Fibrosis Research Center, Birmingham, Alabama
  - Emory Children's Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Solomon GM, Linnemann RW, Rich R, Streby A, Buehler B, Hunter E, Vijaykumar K, Hunt WR, Brewington JJ, Rab A, Bai SP, Westbrook AL, McNicholas-Bevensee C, Hong J, Manfredi C, Barilla C, Suzuki S, Davis BR, Sorscher EJ. Evaluation of elexacaftor-tezacaftor-ivacaftor treatment in individuals with cystic fibrosis and CFTRN1303K in the USA: a prospective, multicentre, open-label, single-arm trial. Lancet Respir Med. 2024 Dec;12(12):947-957. doi: 10.1016/S2213-2600(24)00205-4. Epub 2024 Aug 26. PMID 39208836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at two sites in the United States: The Emory Children's Center in Atlanta, Georgia, and The University of Alabama Cystic Fibrosis Center in Birmingham, Alabama. Participant enrollment began September 4, 2019 and all follow-up assessments were completed by February 13, 2024.
Groups:
- Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency): Substudy 1 - Participants with cystic fibrosis (CF) with evidence of partial function (sweat chloride < 80 milliequivalents per liter (mEq/L) or pancreatic sufficiency) receiving Trikafta for 28 days.
  Trikafta: Participants take Trikafta which is a combination tablet comprised of 100 milligrams (mg) of elexacaftor, 50 mg of tezacaftor and 75 mg of ivacaftor (2 tablets taken in the morning), and 150 mg of ivacaftor taken in the evening.
- Participants Who Encode the N1303K Variant: Substudy 2 - Participants with cystic fibrosis (CF) who encode the N1303K variant receiving Trikafta for 28 days.
  Trikafta: Participants take Trikafta which is a combination tablet comprised of 100 milligrams (mg) of elexacaftor, 50 mg of tezacaftor and 75 mg of ivacaftor (2 tablets taken in the morning), and 150 mg of ivacaftor taken in the evening.
Period: Overall Study
Arm/Group | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency) | Participants Who Encode the N1303K Variant
Started | 22 | 20
Completed | 20 | 20
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency): Participants with cystic fibrosis (CF) with evidence of partial function (sweat chloride < 80 milliequivalents per liter (mEq/L) or pancreatic sufficiency) receiving Trikafta for 28 days.
- Participants Who Encode the N1303K Variant: Participants with cystic fibrosis (CF) who encode the N1303K variant receiving Trikafta for 28 days.
- Total: Total of all reporting groups
Arm/Group | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency) | Participants Who Encode the N1303K Variant | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Customized [Count of Participants; unit: Participants]
  12 to <18 years old | 4 | 8 | 12
  18 or more years old | 18 | 12 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 22 | 18 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Southeast Asian | 2 | 0 | 2
  Black or African American | 3 | 0 | 3
  White or Caucasian | 17 | 18 | 35
  More than one race | 0 | 1 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 20 | 42
CF Medical History [Count of Participants; unit: Participants]
  Pancreatic Insufficiency | 3 | 20 | 23
  CF-related Diabetes | 3 | 4 | 7
  Chronic Sinusitis | 12 | 12 | 24
Percent of Predicted FEV1 [Count of Participants; unit: Participants]
  Less than 50% | 6 | 4 | 10
  50% up to 75% | 4 | 3 | 7
  75% up to 100% | 8 | 13 | 21
  100% or More | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Predicted Forced Expiratory Volume in One Second (FEV1) Among Participants With Evidence of Partial Function
Description: FEV1 provides a direct measurement of patient health among individuals with cystic fibrosis and declines in FEV1 are associated with poor outcomes among those with CF. FEV1 is measured by spirometry and is the maximum amount of air the participant can blow out in one second.
Time Frame: Baseline, Day 28
Population: The Analysis Population includes the intended use population. Two participants with evidence of partial function were found to have cystic fibrosis transmembrane conductance regulator (CFTR) genotypes that were approved by the FDA to use elexacaftor-tezacaftor-ivacaftor while the study was ongoing; these participants were removed from data analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of predicted FEV1
Arm/Group | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency)
Number analyzed (Participants) | 20
percent of predicted FEV1
  Baseline | 74.8 [72.4 to 77.2]
  Day 28 | 76 [73.6 to 78.5]

2. Primary Outcome: Sweat Chloride Among Participants Who Encode the N1303K Variant
Description: Persons with CF have higher levels of chloride in their sweat. Sweat chloride concentrations of less than or equal to 29 mmol/L are considered normal, concentrations of 30-59 mmol/L are considered intermediate and indicate that the individual may have CF. Concentrations of 60 mmol/L and greater mean that a diagnosis of CF is likely.
Time Frame: Baseline, Day 28
Population: The Analysis Population includes the intended use population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/liter
Arm/Group | Participants Who Encode the N1303K Variant
Number analyzed (Participants) | 20
mmol/liter
  Baseline | 109 [105.6 to 112.4]
  Day 28 | 107.9 [104.5 to 111.3]

3. Primary Outcome: Number of Participants With Induced Pluripotent Stem (iPS) Cells Predicting Response to Treatment Among Participants With Evidence of Partial Function
Description: Response of iPS cells (iPSc) to treatment among participants with evidence of partial function was examined to determine whether iPS derived monolayers could predict "personalized" clinical benefit. Cutaneous punch biopsy material was collected from each participant so that iPS cells could be differentiated into airway epithelial monolayers and tested for response to treatment in vitro - as a potential way to predict improvement from Trikafta in vivo.
Time Frame: Baseline
Population: Participants with evidence of partial function were included for the primary outcome measure of examining response of iPS cell derived epithelial monolayers. This analysis includes participants from which samples were successfully obtained, differentiated, and examined using bioelectric measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency)
Number analyzed (Participants) | 8
Participants | 0

4. Secondary Outcome: Percent Predicted Forced Expiratory Volume in One Second (FEV1) Among Participants Who Encode the N1303K Variant
Description: as for outcome 1
Time Frame: Baseline, Day 28
Population: The Analysis Population includes the intended use population.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted FEV1
Arm/Group | Participants Who Encode the N1303K Variant
Number analyzed (Participants) | 20
percent predicted FEV1
  Baseline | 75.8 [73.3 to 78.3]
  Day 28 | 85.3 [82.8 to 87.8]

5. Secondary Outcome: Sweat Chloride Among Participants With Evidence of Partial Function
Description: as for outcome 2
Time Frame: Baseline, Day 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/liter
Arm/Group | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency)
Number analyzed (Participants) | 20
mmol/liter
  Baseline | 66.9 [63.8 to 70.1]
  Day 28 | 57.8 [54.7 to 60.9]

6. Secondary Outcome: Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Domain Score
Description: Participants take the CFQ-R corresponding to their age for assessing quality of life. Responses to questions are coded as 1 = very true or always, 2 = mostly true or often, 3 = somewhat true or sometimes, and 4 = not at all true or never. Some items are reverse scored so that higher scores indicate increased ability and higher quality of life. Scores for items in the respiratory domain are summed and standardized and the standardized score ranges from 1 to 100. A minimum clinically important difference (MCID) of 4 or more points represents improved respiratory-related quality of life.
Time Frame: Baseline, Day 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency) | Participants Who Encode the N1303K Variant
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 66.4 [59.8 to 73.1] | 60.6 [54.6 to 66.5]
  Day 28 | 74.1 [67.5 to 80.7] | 81.4 [75.5 to 87.3]

7. Secondary Outcome: Weight
Description: Weight is measured in kilograms.
Time Frame: Baseline, Day 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency) | Participants Who Encode the N1303K Variant
Number analyzed (Participants) | 20 | 20
kilograms
  Baseline | 75 [74.5 to 75.6] | 57.5 [57.0 to 58.0]
  Day 28 | 75.8 [75.3 to 76.4] | 58.5 [58.0 to 59.1]

8. Secondary Outcome: Body Mass Index (BMI)
Description: Body mass index is calculated as weight in kilograms divided by height in meters squared.
Time Frame: Baseline, Day 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency) | Participants Who Encode the N1303K Variant
Number analyzed (Participants) | 20 | 20
kg/m^2
  Baseline | 25.4 [25.3 to 25.6] | 22.1 [21.9 to 22.3]
  Day 28 | 25.7 [25.5 to 25.9] | 22.5 [22.3 to 22.7]

9. Secondary Outcome: Number of Participants With iPS Cells Predicting Response to Treatment Among Participants Encoding N1303K
Description: Cutaneous punch biopsy material was collected from each participant so that iPS cells could be differentiated into airway epithelial monolayers and tested for response to treatment in vitro - i.e., as a potential way to predict benefit from Trikafta in vivo. By using iPS cells differentiated to exhibit a respiratory epithelial phenotype, the study aims to determine whether iPScs can be used to predict clinical improvement due to Trikafta.
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: Information about adverse events was collected from the time of consent through Day 56.
Arm/Group | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency) | Participants Who Encode the N1303K Variant
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/20
Other Adverse Events (participants affected / at risk) | 17/22 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency) (N=22) | Participants Who Encode the N1303K Variant (N=20)
Hospitalization due to cystic fibrosis pulmonary exacerbation caused by pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Evidence of Partial Function (Sweat Chloride < 80 mEq/L or Pancreatic Sufficiency) (N=22) | Participants Who Encode the N1303K Variant (N=20)
Increased coughing (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Rash (Skin and subcutaneous tissue disorders) | 6 | 0
Increased sputum production (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Diarrhea (Gastrointestinal disorders) | 5 | 0
Fatigue (General disorders) | 4 | 2
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 | 0
Upper respiratory infection (Infections and infestations) | 3 | 4
Body aches (General disorders) | 2 | 2
Increased wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Testicular pain (Reproductive system and breast disorders) | 2 | 0
Headache (General disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eosinophilia (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Decreased forced expiratory volume in one second (FEV1) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decreased appetite (General disorders) | 0 | 1
Coronavirus disease 2019 (COVID-19) (Infections and infestations) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Increased anxiety (Psychiatric disorders) | 0 | 1
Lower respiratory infection (Infections and infestations) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Vision changes (Eye disorders) | 0 | 1
Insomnia (General disorders) | 0 | 1
Dry mouth (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT03506061/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT03506061/ICF_000.pdf